CLINICAL TRIAL: NCT01430455
Title: Tranylcypromine Treatment of Bipolar Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6333
Record Dates: First submitted 2011-09-06; First posted 2011-09-08 (Estimated); Results first posted 2018-03-15 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-02

CONDITIONS: Bipolar Disorder I or II
Keywords: Major Depressive Episode; Depression NOS; Bipolar Disorder; Bipolar Disorder I; Bipolar Disorder II; Bipolar Depression; Major Depression
MeSH Terms: conditions — Depression; Bipolar Disorder; Depressive Disorder, Major | interventions — Tranylcypromine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tranylcypromine (Experimental): Active, open-label tranylcypromine treatment
  Interventions: Drug: Tranylcypromine

INTERVENTIONS:
Drug: Tranylcypromine — Tranylcypromine, between 10 mg/day and 120 mg/day throughout 16 week study
  Other Names: Parnate®

SUMMARY:
This study seeks to investigate whether tranylcypromine (Parnate®) might be an effective treatment of bipolar depression. New treatments are needed, as there is little evidence that standard antidepressants are effective in treating this condition, and the two antipsychotic medications that have indications for bipolar depression can cause substantial side effects. This study will focus specifically on currently depressed outpatients having a bipolar history for whom at least one standard antidepressant medication was ineffective. Patients will be treated openly with tranylcypromine for 8-10 months, depending on treatment response.

ELIGIBILITY:
Inclusion Criteria:

1. History of Bipolar I, II
2. Currently depressed (major depressive episode or depression NOS)
3. Physically healthy or physically stable (i.e.,No changes in medical interventions in past three months or likely for the next three months)
4. On stable and effective mood stabilizer or hypomania deemed sufficiently mild to not require a mood stabilizer.
5. Prior adequate trial on at least one antidepressant.
6. Able to follow a tyramine-free diet
7. Must speak English

Exclusion Criteria:

1. Current psychosis
2. past psychosis not occurring during an episode of mania or depression
3. prior nonremission to tranylcypromine 60 mg/d (or greater)
4. currently taking effective medication precluded while taking a Monoamine Oxidase Inhibitor (e.g., a psychostimulant or a serotonin re-uptake inhibitor)
5. current (last six months) drug or alcohol abuse or dependence
6. significant suicide risk
7. significant cardiovascular risk

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2014-02 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- See also: Depression Evaluation Service — http://depression-nyc.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tranylcypromine
Started | 7
Completed | 5
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Switched to follow-up phase | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tranylcypromine
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: 29 Item Hamilton Rating Scale for Depression (HamD29)
Description: 29 Item Hamilton Rating Scale for Depression (HamD29) is the 29 item version of the most common depression rating scale. The scores represented here are the average scores at baseline and after 16 weeks of open label treatment. The scale is rated from 0-89 with higher scores representing a more depressed state.
Time Frame: Hamilton 29 score at baseline (start date of medication) and week 16
Population: 2 patients who did not make it to week 16 (one dropped out at week 3 and one dropped out at week 9)
Measure: Mean (Standard Error); unit: Hamilton Depression score
Arm/Group | Tranylcypromine
Number analyzed (Participants) | 7
Hamilton Depression score
  Baseline Score | 27.0 (1.4)
  Week 16 Score: number analyzed (Participants) | 5
  Week 16 Score | 5.8 (2.1)

ADVERSE EVENTS:
Arm/Group | Tranylcypromine
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 6/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tranylcypromine (N=7)
Lightheadedness (Vascular disorders) | 2 (2)
Weight gain (Metabolism and nutrition disorders) | 1 (1)
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)
increased appetite (Metabolism and nutrition disorders) | 1 (1)
Light Sensitivity (Eye disorders) | 1 (1)
muscle tension (Musculoskeletal and connective tissue disorders) | 1 (1)
water retention (General disorders) | 1 (2)
postural hypotension (Vascular disorders) | 1 (2)
insomnia (Nervous system disorders) | 1 (1)
constipation (Gastrointestinal disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Leg cramps (Musculoskeletal and connective tissue disorders) | 1 (1)
Mild ataxia (General disorders) | 2 (3)
Dry Mouth (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No